CLINICAL TRIAL: NCT03904355
Title: Effects of Intramural Fibroids That do Not Distort the Uterine Cavity on IVF Outcome
Brief Title: Effects of Intramural Fibroids on IVF Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 54
Record Dates: First submitted 2019-03-31; First posted 2019-04-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Infertility, Female; Assisted Reproduction
MeSH Terms: conditions — Infertility, Female | interventions — Gonadotropins; Ovulation Induction; Chorionic Gonadotropin; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiboroid group (Active Comparator): Women with intramural myoma no reaching the cavity
  Interventions: Drug: Gonadotropins; Drug: human chorionic gonadotropin; Procedure: Ovum pick up; Procedure: Embryo transfer
- Non fibroid group (Active Comparator): Women without myomas
  Interventions: Drug: Gonadotropins; Drug: human chorionic gonadotropin; Procedure: Ovum pick up; Procedure: Embryo transfer

INTERVENTIONS:
Drug: Gonadotropins — Gonadotropin stimulation of follicular growth
  Other Names: Ovarian stimulation
Drug: human chorionic gonadotropin — HCG triggering of ovulation
  Other Names: Triggering of ovulation
Procedure: Ovum pick up — 34 to 36 hours after oocyte retrieval
Procedure: Embryo transfer — Transfer of 2 grade 1 embryo on day 2,3 or 5 from oocyte retrieval

SUMMARY:
A cohort study involving 200 women candidate for IVF / ICSI cycles . The participants will be assessed through full history-taking with special consideration to age and the duration, type, and cause of infertility. The medical examination included general, abdominal, and vaginal examinations. Finally, an ultrasonography examination was performed to check for the presence of three or more preantral follicles and to exclude ovarian cysts.

On day 3 of a natural cycle, a baseline levels of FSH, luteinizing hormone (LH),

, estradiol and anti-Müllerian hormone (AMH).Ovarian stimulation was performed using a long, antagonist, or short protocol. They were assigned to one of the 2 groups according to having an intramural myoma not indenting the cavity or not. All will be followed up by transvaginal ultrasonography . When two or more follicles had reached a mean diameter of 18 mm, oocyte maturation was triggered by intramuscular administration of hCG. Embryo transfer will be done at day 2, 3 or 5 according to the circumstances.

DETAILED DESCRIPTION:
A cohort study involving 200 women candidate for IVF / ICSI cycles . The participants will be assessed through full history-taking with special consideration to age and the duration, type, and cause of infertility. The medical examination included general, abdominal, and vaginal examinations. Finally, an ultrasonography examination was performed to check for the presence of three or more preantral follicles and to exclude ovarian cysts.

On day 3 of a natural cycle, a baseline levels of FSH, luteinizing hormone (LH),

, estradiol and anti-Müllerian hormone (AMH).Ovarian stimulation was performed using a long, antagonist, or short protocol. They were assigned to one of the 2 groups according to having an intramural myoma not indenting the cavity or not. All will be followed up by transvaginal ultrasonography . When two or more follicles had reached a mean diameter of 18 mm, oocyte maturation was triggered by intramuscular administration of hCG. Embryo transfer will be done at day 2, 3 or 5 according to the circumstances.

ELIGIBILITY:
Inclusion Criteria:

* age younger than 40 years
* FSH) less than 10 IU/L
* serum prolactin level normal
* uterine cavity abnormality was excluded by hysteroscopy or hysterosalpingography.

Exclusion Criteria:

* abnormal endocrine function (e.g. abnormal thyroid or adrenal function)
* ovarian cysts,
* hydrosalpinx
* endometrial polyps
* male partner with azoospermia
* ICSI performed for preimplantation genetic diagnosis.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  appearance of one or more intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided